CLINICAL TRIAL: NCT04945746
Title: Study Evaluating the Prioritization of Ablation Zones According to the Stability of the Dispersion
Brief Title: Dispersion Stability
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSJ_Dispersion Stability_2021
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Software VX1 + Stability (Experimental): Utilization of the software VX1 + Stability
  Interventions: Procedure: AF ablation

INTERVENTIONS:
Procedure: AF ablation — AF ablation using the Volta Medical VX1 CE marked software and a new criteria to establish a priority of the dispersed zones according to the stability of the core algorithm's response (thanks to the new software module under study named "stability").

SUMMARY:
To assess the acute efficacy of ablation of the most stable VX1 areas (levels 2 and 3) in terms of the rate of acute AF termination.

Identify the spatial distribution of dispersion stability levels based on VX1. Document the rate of adverse events. To assess the long-term efficacy of ablation of the most stable VX1 areas in terms of the absence of documented arrhythmias during a 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older candidates with Persistent or long-standing persistent AF with documentation of (ECG, Holter, physician's letter):

   * AF duration of ≥ 3 months and ≤ 5 years or
   * 1 effective cardioversion followed by AF recurrence lasting ≥ 3 months
2. Continuous anticoagulation with warfarin (INR 2-3) or NOAC for > 4 weeks prior to ablation
3. Patients must be able and willing to provide written informed consent to participate in the clinical trial
4. Maximum of 50% of patients (13 patients) in persistent AF < 12 months (>30% of long-standing persistent AF ≥ 12 months)
5. Being affiliated to a social security scheme or beneficiary of such a scheme

Exclusion Criteria:

1. Paroxysmal and short-standing persistent AF < 3 months
2. Severe obesity (BMI > 45)
3. LA thrombus on Transesophageal Echocardiography (TEE) prior to procedure
4. Contraindications to anticoagulation (heparin, warfarin or NOAC)
5. Patients who are or may potentially be pregnant
6. Any cardiac surgery within the past 2 months (60 days) (includes PCI)
7. Myocardial infarction within the past 2 months (60 days)
8. History of blood clotting or bleeding abnormalities
9. Documented thromboembolic event (including TIA) within the past 12 months (365 days)
10. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months (365 days)
11. Unstable angina within the past month
12. Acute illness or active systemic infection or sepsis (including COVID 19)
13. Enrollment in an investigational study evaluating another device, biologic, or drug
14. Presence of intramural thrombus, tumor or other abnormality or condition that precludes vascular access, or manipulation of the catheter
15. Life expectancy or other disease processes likely to limit survival to less than 12 monthsLife expectancy or other disease processes likely to limit survival to less than 12 months
16. Acute Covid-19 infection (fever and/or biological inflammatory syndrome, and positive test documented)
17. Patient protected (guardianship or curatorship), or deprived of liberty by a judicial or administrative decision;
18. Person subject to a safeguard measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2025-01-28 (Estimated)

PRIMARY OUTCOMES:
AF termination rate after ablation of the most stable regions (levels 3 and 2) | at the end of the procedure
  sinus rhythm at the end of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Joseph Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No